CLINICAL TRIAL: NCT02897050
Title: Phase II Trial of Neoadjuvant Docetaxel ± Metronomic Capecitabine/CTX Followed by FEC in Women With Operable Triple Negative Breast Cancer
Brief Title: Trial of Neoadjuvant Docetaxel ± Metronomic Capecitabine/CTX Followed by FEC in Women With Operable Triple Negative Breast Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., President of Sun Yat-sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCCT2016001
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine; Cyclophosphamide; Tablets; Fluorouracil; Epirubicin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T+mCX followed by FEC (Experimental): Docetaxel 75mg/m2, iv, d1 + CTX 50 mg/d, po, d1-d21 + capecitabine 1200mg/m2/d, po, d1-d21 * 3 cycles (21 days per cycle) followed by fluorouracil 500mg/m2,iv,d1 + epirubicin 100mg/m2,iv,d1 + cyclophosphamide 500mg/m2,iv,d1 * 3 cycles (21 days per cycle)
  Interventions: Drug: Docetaxel; Drug: Capecitabine; Drug: Cyclophosphamide (tablet); Drug: Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide (injection)
- T followed by FEC (Active Comparator): Docetaxel 100mg/m2, iv, d1 * 3 cycles (21 days per cycle) followed by fluorouracil 500mg/m2,iv,d1 + epirubicin 100mg/m2,iv,d1 + cyclophosphamide 500mg/m2,iv,d1 * 3 cycles (21 days per cycle)
  Interventions: Drug: Docetaxel; Drug: Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide (injection)

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75mg/m2, iv, d1 or 100mg/m2, iv, d1
Drug: Capecitabine — Capecitabine 1200mg/m2/d, po, d1-d21
  Other Names: Xeloda
  Arms: T+mCX followed by FEC
Drug: Cyclophosphamide (tablet) — Cyclophosphamide 50 mg/d, po, d1-d21
  Other Names: CTX
  Arms: T+mCX followed by FEC
Drug: Fluorouracil — Fluorouracil 500mg/m2, iv, d1
  Other Names: 5-Fu
Drug: Epirubicin — Epirubicin 100mg/m2, iv, d1
Drug: Cyclophosphamide (injection) — Cyclophosphamide 500mg/m2, iv, d1
  Other Names: CTX

SUMMARY:
This multi-center, open-label, phase II randomized controlled trial is to evaluate the efficacy of docetaxel(T) combined with metronomic cyclophosphamide/capecitabine (mCX) followed by fluorouracil /epirubicin/cyclophosphamide (FEC) versus T followed by FEC as neoadjuvant chemotherapy in treating women with triple negative breast cancer (TNBC), and to study the anti-tumor immune effect of metronomic neoadjuvant chemotherapy. 186 stage M0 TNBC patients who had a primary tumor > 2cm by imaging or an axillary lymph node > 2cm by imaging are randomly enrolled to receive neoadjuvant T combined with mCX (3 cycles) followed by FEC (3 cycles) or T (3cycles) followed by FEC (3 cycles) before surgery. The primary end point is pathological complete response (pCR) rate, and the secondary end points include: clinical response rate, toxicities, breast-conserving rate, Ki67 and CD31 reduction rate, changes in the percentages of peripheral blood or tumor microenvironmental regulatory T cells (Treg), T helper cells (Th), CD8+ T cell, and tumor-specific CTL, and changes in tumor microenvironmental immune cytokines. Once there is a significant statistical difference in terms of pCR rate between two groups, 3-year disease-free survival (DFS) and 3-year overall survival (OS) will be included in the secondary end points. The aims of this study are to determine whether the neoadjuvant T combined with metronomic CX followed by FEC can significantly increase the pCR rate in TNBC with acceptable toxicity, and to explore the anti-tumor immune effect of metronomic neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* The patients signed the written informed consent
* The patients present with non-metastatic unilateral invasive ER-negative (IHC<10%), PR-negative(IHC<10%), HER2-negative breast cancer with a primary breast tumor > 2cm by imaging or an axillary lymph node > 2cm by imaging.
* 18 years old< age < 70 years old.
* The patients have no history of hormone therapy, chemotherapy, breast cancer surgery and radiotherapy.
* The patients have normal cardiac functions by echocardiography.
* The patients' ECOG scores are ≤2.
* The patients can swallow pills.
* The results of patients' blood tests are as follows:

  * Hb≥90g/L;
  * WBC≥4E+9/L;
  * Plt≥100E+9/L;
  * Neutrophils≥1.5E+9/L;
  * ALT and AST ≤ triple of normal upper limit;
  * TBIL ≤ 1.5 times of normal upper limit;
  * Creatinine ≤ 1.5 times of normal upper limit.

Exclusion Criteria:

* The patients have other cancers at the same time or have the history of other cancers except controlled skin basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of cervix uterus;
* The patients have active infections that were not suitable for chemotherapy;
* The patients have severe non-cancerous diseases.
* The patients have bilateral breast cancers or male breast cancers or inflammatory breast cancers.
* The patients are undergoing current administration of anti-cancer therapies, or are attending other clinical trials.
* The patients are in some special conditions that they cannot understand the written informed consent, such as they are demented or hawkish.
* The patients have allergic history or contraindication of any of the interventional drugs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | at definitive surgery (20-24 weeks after the first dose of study medication)

SECONDARY OUTCOMES:
Ultrasound response rate | at definitive surgery (20-24 weeks after the first dose of study medication)
Breast-conserving surgery rate | at definitive surgery (20-24 weeks after the first dose of study medication)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | during on-neoadjuvant therapy period (defined as the period from the first dose of study medication up to 30 days of the last dose)
Tumor Ki67 reduction rate in relation to neoadjuvant therapy | at definitive surgery (20-24 weeks after the first dose of study medication)
Tumor CD31 reduction rate in relation to neoadjuvant therapy | at definitive surgery (20-24 weeks after the first dose of study medication)
Peripheral blood CD8+ T cell percentage change in relation to neoadjuvant therapy | at definitive surgery (20-24 weeks after the first dose of study medication)
Peripheral blood regulatory T cell percentage change in relation to neoadjuvant therapy | at definitive surgery (20-24 weeks after the first dose of study medication)
Peripheral blood tumor specific T cell (CTL) percentage change in relation to neoadjuvant therapy | at definitive surgery (20-24 weeks after the first dose of study medication)
Peripheral blood T helper cell percentage change in relation to neoadjuvant therapy | at definitive surgery (20-24 weeks after the first dose of study medication)

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xinjiang Medical School Cancer Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided